CLINICAL TRIAL: NCT02712827
Title: A Randomized Controlled Trial Comparing Short Term Outcomes of Self-gripping (Progrip) Mesh With Fibrin Glue Mesh Fixation in Laparoscopic Total Extraperitoneal (TEP) Inguinal Hernia Repair
Brief Title: Comparison of Different Meshes in Laparoscopic Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Dominic C.C. Foo, Clinical Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UW 16-042
Record Dates: First submitted 2016-03-10; First posted 2016-03-18 (Estimated); Last update posted 2018-11-27 (Actual); Status verified 2018-11

CONDITIONS: Hernia, Inguinal
Keywords: self-gripping mesh, fibrin glue, total extraperitoneal
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Progrip (Experimental): The Progrip group is the intervention group. Patients will undergo laparoscopic total extraperitoneal repair of inguinal hernia. The surgeon will use a self-gripping mesh to repair the hernia. No fixation is required for the mesh.
  Interventions: Procedure: Progrip
- Non-Progrip (Active Comparator): The Non-Progrip group is the control group.
  Operation is performed under general anesthesia. A standard three-trocar technique is used: one infra-umbilical camera trocar (1cm) and two 5mm trocars placed at midline between the umbilicus and pubic bone (or one at the side of inguinal hernia). A laparoscope is inserted to the preperitoneal space through the incision. The space is insufflated with carbon dioxide. Dissection is performed, hernia content (if any) is reduced.
  A non self-gripping synthetic mesh is placed. Fibrin glue is used for fixation.
  Interventions: Procedure: Non-Progrip

INTERVENTIONS:
Procedure: Progrip — Self-fixating mesh
  Arms: Progrip
Procedure: Non-Progrip — Non self-fixating mesh with the use of glue
  Arms: Non-Progrip

SUMMARY:
The placement of mesh is important in hernia surgery as it helps to reduce recurrence, yet the method of fixation of mesh may cause pain after surgery. In laparoscopic hernia repair, surgeon uses different methods to fix the mesh in large hernia defects or bilateral inguinal hernias. Progrip is a special mesh developed by manufacturer that it can be self-gripped to tissue, as a result no fixation is required after placement. There are few data about Progrip in laparoscopic hernia repair. In this randomized controlled trial we would like to compare the use of Progrip with the "conventional" mesh in laparoscopic hernia repair. Surgery is performed in the usual manner; prior to placement of mesh, surgeon will get the randomization result for that particular patient: Progrip and non-Progrip group. No fixation is required for Progrip group, while fixation with fibrin glue is needed for non-Progrip group. Intraoperative data (e.g. mesh deployment time, operative time, etc) will be collected. Patients will be assessed in clinic at 2-week, 3-month, 6-month and 1-year interval after surgery. Additional visits may be arranged if considered necessary. At follow up patient will be seen by surgeon first to review the wound condition and to look for any recurrence; while other post-operative data including total analgesic usage (number of tablets), return to normal activities (days), return to work (days), pain score etc will be assessed and recorded by a trained nurse who is blinded to the treatment that patient received. Any hernia recurrence will be recorded and treated accordingly. Primary aim of this study is to look for any difference of the 2 groups in terms of postoperative pain and quality of life scores.

DETAILED DESCRIPTION:
Inguinal hernia repair is one of the common surgeries performed by general surgeon all over the world. Tension-free Lichtenstein repair is the most common technique used in open repair, while many surgeons perform laparoscopic hernia repair: total extraperitoneal repair (TEP) and transabdominal preperitoneal repair (TAPP). Laparoscopic surgery is considered to reduce postoperative pain, the incidence of wound complications and time to return to activities of daily living. Both techniques are based on the principle of tension free repair and rely on mesh placement in the preperitoneal space to exclude the inguinal defect and reinforce the abdominal wall; the recurrence rate following tension-free hernia repair is reported to be low and in the range of 1-4%.

Chronic pain after an inguinal hernia repair is a well recognized complication, irrespective of technique. The incidence of chronic pain is estimated to be around 5-10%. Many factors contributed to the development of chronic pain, and one of the factors being the type of mesh fixation method. Common types of mesh fixation methods in laparoscopic hernia repair are traumatic fixation - the use of tacks (absorbable or non-absorbable) or atraumatic fixation, e.g. the use of fibrin glue; while some surgeons do not fix the mesh. No fixation is practiced by some surgeons in unilateral repair as some studies showed that there was no difference in recurrence rate and incidence of chronic pain between fixation or no fixation groups, yet in these studies hernia opening was small (<3cm) or not measured. It is generally agreed that fixation is indicated in large hernias (defect size >3cm), bilateral hernias and recurrent hernias in order to avoid early mesh dislocation and hernia recurrence.

Study has shown that the use of tacks caused more early postoperative pain. Manufacturers try to develop self-gripping mesh with the aim to reduce chronic pain. ProgripTM (Covidien) is a lightweight, self-gripping mesh composed of monofilament polyester and polylactic acid (PLA) microgrips indicated for inguinal hernia repair. The resorbable microgrips provide immediate adherence to surrounding muscle and adipose tissue during hernia surgery, as a result no fixation method is required. Studies have shown that ProgripTM is associated with less pain in the early recovery period when used in open Lichtenstein repair, yet there are few studies of ProgripTM in laparoscopic hernia repair.

In Hong Kong, TEP is the preferred approach for most surgeons who perform laparoscopic hernia surgery. In this trial, patients with inguinal hernia who is suitable for TEP are recruited. TEP will be performed in the usual manner. Surgeon will assess the size of hernia defect prior to mesh insertion. For patients with large hernia defect or bilateral inguinal hernia that required mesh fixation, they will be randomized in two groups: ProgripTM and non-ProgripTM group. For ProgripTM no addition fixation is necessary, while for non-ProgripTM fixation is indicated. As tacks are known to be associated with postoperative pain, fibrin glue is designated as the fixation method in non- ProgripTM group in this study.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18
* Unilateral inguinal hernia with large hernia defect size (>3cm)
* Bilateral inguinal hernias
* American Society of Anesthesiologists (ASA) score: 1-2
* Provision of written informed consent

Exclusion Criteria:

* Any prior surgery for ipsilateral inguinal hernia (i.e. recurrent inguinal hernia)
* American Society of Anesthesiologists (ASA) score: 3 or above
* History of major abdominal surgery that may result in difficulty in development of preperitoneal space
* Subject is pregnant or breast feeding
* Any serious concomitant illness with short life expectancy
* Subject who is not able to attend follow up postoperatively

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Chronic pain | 3 months post surgery
  Chronic pain after hernia surgery was defined as the presence of pain at rest at the groin area. The severity of pain will be measured by a linear analogue pain score sacle from 0 to 10. Score >= 1 indicate the presence of pain.

SECONDARY OUTCOMES:
mesh deployment time | 1 day
  the time for mesh deployment during surgery
intraoperative complications | 1 day
  intraoperative complications
hernia recurrence rate | 1 year
  hernia recurrence rate
quality of life | 1 year
  quality of life scores

CONTACTS AND LOCATIONS:
Overall Officials: Dominic, Chi Chung Foo, MBBS, Principal Investigator — The University of Hong Kong
Locations (1):
- Tung Wah Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bresnahan E, Bates A, Wu A, Reiner M, Jacob B. The use of self-gripping (Progrip) mesh during laparoscopic total extraperitoneal (TEP) inguinal hernia repair: a prospective feasibility and long-term outcomes study. Surg Endosc. 2015 Sep;29(9):2690-6. doi: 10.1007/s00464-014-3991-y. Epub 2014 Dec 18. PMID 25519425
- [Background] Kingsnorth A, Gingell-Littlejohn M, Nienhuijs S, Schule S, Appel P, Ziprin P, Eklund A, Miserez M, Smeds S. Randomized controlled multicenter international clinical trial of self-gripping Parietex ProGrip polyester mesh versus lightweight polypropylene mesh in open inguinal hernia repair: interim results at 3 months. Hernia. 2012 Jun;16(3):287-94. doi: 10.1007/s10029-012-0900-y. Epub 2012 Mar 28. PMID 22453675
- [Background] Teng YJ, Pan SM, Liu YL, Yang KH, Zhang YC, Tian JH, Han JX. A meta-analysis of randomized controlled trials of fixation versus nonfixation of mesh in laparoscopic total extraperitoneal inguinal hernia repair. Surg Endosc. 2011 Sep;25(9):2849-58. doi: 10.1007/s00464-011-1668-3. Epub 2011 Apr 13. PMID 21487873
- [Background] Tam KW, Liang HH, Chai CY. Outcomes of staple fixation of mesh versus nonfixation in laparoscopic total extraperitoneal inguinal repair: a meta-analysis of randomized controlled trials. World J Surg. 2010 Dec;34(12):3065-74. doi: 10.1007/s00268-010-0760-5. PMID 20714896
- [Background] Belyansky I, Tsirline VB, Klima DA, Walters AL, Lincourt AE, Heniford TB. Prospective, comparative study of postoperative quality of life in TEP, TAPP, and modified Lichtenstein repairs. Ann Surg. 2011 Nov;254(5):709-14; discussion 714-5. doi: 10.1097/SLA.0b013e3182359d07. PMID 21997807
- [Background] Simons MP, Aufenacker T, Bay-Nielsen M, Bouillot JL, Campanelli G, Conze J, de Lange D, Fortelny R, Heikkinen T, Kingsnorth A, Kukleta J, Morales-Conde S, Nordin P, Schumpelick V, Smedberg S, Smietanski M, Weber G, Miserez M. European Hernia Society guidelines on the treatment of inguinal hernia in adult patients. Hernia. 2009 Aug;13(4):343-403. doi: 10.1007/s10029-009-0529-7. Epub 2009 Jul 28. PMID 19636493
- [Background] Pokorny H, Klingler A, Schmid T, Fortelny R, Hollinsky C, Kawji R, Steiner E, Pernthaler H, Fugger R, Scheyer M. Recurrence and complications after laparoscopic versus open inguinal hernia repair: results of a prospective randomized multicenter trial. Hernia. 2008 Aug;12(4):385-9. doi: 10.1007/s10029-008-0357-1. Epub 2008 Feb 19. PMID 18283518
- [Background] Myers E, Browne KM, Kavanagh DO, Hurley M. Laparoscopic (TEP) versus Lichtenstein inguinal hernia repair: a comparison of quality-of-life outcomes. World J Surg. 2010 Dec;34(12):3059-64. doi: 10.1007/s00268-010-0730-y. PMID 20703474
- [Background] Langeveld HR, van't Riet M, Weidema WF, Stassen LP, Steyerberg EW, Lange J, Bonjer HJ, Jeekel J. Total extraperitoneal inguinal hernia repair compared with Lichtenstein (the LEVEL-Trial): a randomized controlled trial. Ann Surg. 2010 May;251(5):819-24. doi: 10.1097/SLA.0b013e3181d96c32. PMID 20395851
- [Background] Eklund AS, Montgomery AK, Rasmussen IC, Sandbue RP, Bergkvist LA, Rudberg CR. Low recurrence rate after laparoscopic (TEP) and open (Lichtenstein) inguinal hernia repair: a randomized, multicenter trial with 5-year follow-up. Ann Surg. 2009 Jan;249(1):33-8. doi: 10.1097/SLA.0b013e31819255d0. PMID 19106673
- [Background] Dulucq JL, Wintringer P, Mahajna A. Laparoscopic totally extraperitoneal inguinal hernia repair: lessons learned from 3,100 hernia repairs over 15 years. Surg Endosc. 2009 Mar;23(3):482-6. doi: 10.1007/s00464-008-0118-3. Epub 2008 Sep 23. PMID 18810548
- [Background] Gong K, Zhang N, Lu Y, Zhu B, Zhang Z, Du D, Zhao X, Jiang H. Comparison of the open tension-free mesh-plug, transabdominal preperitoneal (TAPP), and totally extraperitoneal (TEP) laparoscopic techniques for primary unilateral inguinal hernia repair: a prospective randomized controlled trial. Surg Endosc. 2011 Jan;25(1):234-9. doi: 10.1007/s00464-010-1165-0. Epub 2010 Jun 15. PMID 20552368
- [Background] Rutkow IM. Demographic and socioeconomic aspects of hernia repair in the United States in 2003. Surg Clin North Am. 2003 Oct;83(5):1045-51, v-vi. doi: 10.1016/S0039-6109(03)00132-4. PMID 14533902